CLINICAL TRIAL: NCT02334449
Title: A First-in-human, Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Oral Dose Study, to Assess the Safety, Tolerability and Pharmacokinetics of LML134 in Healthy Volunteers
Brief Title: First-in-human Study to Assess the Safety and Pharmacokinetics of LML134 in Healthy Volunteers
Acronym: LML134
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLML134X2101; 2014-000937-22 (EudraCT Number)
Record Dates: First submitted 2014-11-14; First posted 2015-01-08 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Healthy Volunteers
Keywords: healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single dose study part (Experimental): there will be 8 cohorts of healthy volunteers dosed with single doses of LML134 (8 planned dose levels) or with placebo and 2 potential additional cohorts (also dosed with single dose of LML134 or placebo)
  Interventions: Drug: LML134; Drug: Placebo
- Multiple dose study part (Experimental): there will be 3 cohorts of healthy volunteers dosed with multiple doses of LML134 (3 planned dose levels) or placebo and one potential additional cohort (also dosed with multiple doses of LML134 or placebo)
  Interventions: Drug: LML134; Drug: Placebo

INTERVENTIONS:
Drug: LML134 — LML134 will be administered first as single doses and then as multiple doses
Drug: Placebo — All study cohorts (except food effect cohort) are placebo controlled

SUMMARY:
Phase I study to assess the safety, tolerability and pharmacokinetics of ascending single and multiple doses of the investigational medicinal product in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects age 18 to 55 years of age included, and in good health as determined by medical history, physical examination, vital signs, electrocardiogram, and laboratory tests.
* Written informed consent must be obtained before any assessment is performed.
* Able to communicate well with the Investigator, to understand and comply with the requirements of the study.

Exclusion Criteria:

* History or presence of epilepsy or of seizures or convulsions of any kind.
* Any clinically relevant abnormalities identified in the resting EEG during screening, or pre-ictal signs or other clinically relevant abnormalities in the hyperventilation or intermittent photic stimulation EEG during screening.
* History of head trauma leading to clinically significant symptoms in the past two years.
* Applies only to subjects enrolled in Part 2 MAD. Score "yes" on item 4 or item 5 of the Suicidal Ideation section of the C-SSRS, if this ideation occurred in the past 6 months, or "yes" on any item of the Suicidal Behavior section, except for the "Non-Suicidal Self-Injurious Behavior" (item also included in the Suicidal Behavior section), if this behavior occurred in the past 2 years.
* Significant illness including any clinically significant infectious disease which has not resolved within two (2) weeks prior to initial dosing.
* History or presence of significant hematological abnormalities or immunodeficiency or any condition that might compromise the immune system (infection, vaccination), of any etiology as indicated by clinically significantly abnormal values of any of the following hematologic parameters: thrombocyte, RBC count, total WBC count and differentials presented as % of total white blood cell count and as absolute concentrations.
* History or presence of any thyroid disease as indicated by any clinically relevant abnormality on thyroid stimulating hormone test (TSH).
* History or presence of any chronic eye disease other than refractive error, strabismic amblyopia, or anisometropic amblyopia.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Adverse events assessments after single and multiple ascending dose administration at baseline and repeatedly until study completion | Starting about 24 hours before dosing and continued until about 7-14 days after last dose
  This safety outcome combines the measure of the number of subjects experiencing adverse events (AEs), the nature and severity of those AEs and their relationship to the study treatments.
Cardiovascular safety assessments after single and multiple ascending dose administration at baseline and repeatedly until study completion | Starting about 24 hours before dosing and continued until about 7-14 days after last dose
  This safety outcome combines the measure of a set of cardiovascular safety parameters extracted from ECGs, 25 hours-Holter ECGs and from vital signs assessments
Central nervous system safety assessments after single and multiple ascending dose administration at baseline and repeatedly until study completion | Starting about 24 hours before dosing and continued until about 7-14 days after last dose
  This safety outcome combines the measure of a set of central nervous system safety parameters extracted from EEGs and neurological examinations
Ocular safety assessments after single and multiple ascending dose administration at baseline and repeatedly until study completion | Starting about 24 hours before dosing and continued until about 7-14 days after last dose
  This safety outcome combined the measure of a set of ocular parameters including best corrected visual acuity and other parameters assessed by the mean of slit lamp biomicroscopy and dilated ophthalmoscopy examinations and by optical coherence tomography and electroretinography
General safety assessments after single and multiple ascending dose administration at baseline and repeatedly until study completion | Starting about 24 hours before dosing and continued until about 7-14 days after last dose
  This general safety outcome combines the measure of blood laboratory parameters and the outcome of physical examinations

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of LML134: time to reach the maximum concentration after a single drug administration (Tmax) in Part 1 and in Part 3 | Starting 1hour prior to dosing on Day 1 and until 72 hours after dosing (Day 4)
  Serum samples will be collected on Day 1: 1hr predose; 0,25h; 0,5h; 1h; 1,5h; 2h; 3h; 4h; 6h; 8h; 12h; 16h post dose, on Day 2: 24h and 36h post dose, on Day 3: 48h and 60h post dose and on Day 4: 72h post dose. This outcome measure shows the mean of all subject values resulting from each time point specified above, in Parts 1 and 3.
  In Part 3, the outcome measure is done once without food intake and once after the intake of a high fat breakfast (in 2 different periods). Both outcomes (with and without breakfast intake) will be compared to assess the effect of a high fast breakfast on LML134 Tmax
PK of LML134: Observed maximum serum concentration following single drug administration (Cmax) in Part 1 and Part 3 | Starting 1hour prior to dosing on Day 1 and until 72 hours after dosing (Day 4)
  Serum samples will be collected on Day 1: 1hr predose; 0,25h; 0,5h; 1h; 1,5h; 2h; 3h; 4h; 6h; 8h; 12h; 16h post dose, on Day 2: 24h and 36h post dose, on Day 3: 48h and 60h post dose and on Day 4: 72h post dose. This outcome measure shows the mean of all subject values resulting from each time point specified above, in Parts 1 and 3.
  In Part 3, the outcome measure is done once without food intake and once after the intake of a high fat breakfast (in 2 different periods). Both outcomes (with and without breakfast intake) will be compared to assess the effect of a high fast breakfast on LML134 Cmax.
PK of LML134: Area under the serum concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) in Part 1 and Part 3 | Starting 1hour prior to dosing on Day 1 and until 72 hours after dosing (Day 4)
  Serum samples will be collected on Day 1: 1hr predose; 0,25h; 0,5h; 1h; 1,5h; 2h; 3h; 4h; 6h; 8h; 12h; 16h post dose, on Day 2: 24h and 36h post dose, on Day 3: 48h and 60h post dose and on Day 4: 72h post dose. This outcome measure shows the mean of all subject values resulting from each time point specified above, in Parts 1 and 3. In Part 3, the outcome measure is done once without food intake and once after the intake of a high fat breakfast (in 2 different periods). Both outcomes (with and without breakfast intake) will be compared to assess the effect of a high fast breakfast on LML134 AUClast.
PK of LML134: time to reach the maximum concentration after the first drug administration (Tmax) in Part 2 | Starting 1hour prior the first dose administration (Day 1) until 24hr after the first dose administration on Day 2
  Serum samples will be collected on Day 1: 1hr predose; 0,25h; 0,5h; 1h; 1,5h; 2h; 3h; 4h; 6h; 8h; 12h; 16h post dose and on Day 2: 24h post dose. This outcome measure shows the mean of all subject values resulting from each time point specified above.
PK of LML134: time to reach the maximum concentration after the last drug administration (Tmax) in Part 2 | Starting 1hour prior the first dose administration (Day 1) until 48hour after the last dose administration (Day 17)
  Serum samples will be collected on Day 1: 1hr predose; 0,25h; 0,5h; 1h; 1,5h; 2h; 3h; 4h; 6h; 8h; 12h; 16h post dose, on Day 2: 24h post dose, on Day 3: 1hr prior the second dose administration, on Days 4, 5, 6, 8, 10, 12, 13, 14: 1hr prior dosing, on Day 15 (last time the drug is administered): 1hr predose; 0,25h; 0,5h; 1h; 1,5h; 2h; 3h; 4h; 6h; 8h; 12h; 16h post dose, on Day 16: 24h post dose and Day 17: 48h post dose. This outcome measure shows the mean of all subject values resulting from each time point specified above.
PK of LML134: Observed maximum serum concentration following the first drug administration (Cmax) in Part 2 | Starting 1hour prior the first dose administration (Day 1) until 24hr after the first dose administration on Day 2
  Serum samples will be collected on Day 1: 1hr predose; 0,25h; 0,5h; 1h; 1,5h; 2h; 3h; 4h; 6h; 8h; 12h; 16h post dose and on Day 2: 24h post dose. This outcome measure shows the mean of all subject values resulting from each time point specified above.
PK of LML134: Observed maximum serum concentration following drug administration at steady state (Cmax,ss) in Part 2 | Starting 1hour prior the first dose administration (Day 1) until 48hour after the last dose administration (Day 17)
  Serum samples will be collected on Day 1: 1hr predose; 0,25h; 0,5h; 1h; 1,5h; 2h; 3h; 4h; 6h; 8h; 12h; 16h post dose, on Day 2: 24h post dose, on Day 3: 1hr prior the second dose administration, on Days 4, 5, 6, 8, 10, 12, 13, 14: 1hr prior dosing, on Day 15 (last time the drug is administered): 1hr predose; 0,25h; 0,5h; 1h; 1,5h; 2h; 3h; 4h; 6h; 8h; 12h; 16h post dose, on Day 16: 24h post dose and Day 17: 48h post dose. This outcome measure shows the mean of all subject values resulting from each time point specified above.
PK of LML134: Area under the serum concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) after the first dose administration in Part 2 | Starting 1hour prior the first dose administration (Day 1) until 24hr after the first dose administration on Day 2
  Serum samples will be collected on Day 1: 1hr predose; 0,25h; 0,5h; 1h; 1,5h; 2h; 3h; 4h; 6h; 8h; 12h; 16h post dose and on Day 2: 24h post dose. This outcome measure shows the mean of all subject values resulting from each time point specified above.
PK of LML134: The area under the serum concentration-time curve from time zero to the end of the dosing interval tau at steady state (AUCtau,ss) in Part 2 | Starting 1hour prior the first dose administration (Day 1) until 48hour after the last dose administration (Day 17)
  Serum samples will be collected on Day 1: 1hr predose; 0,25h; 0,5h; 1h; 1,5h; 2h; 3h; 4h; 6h; 8h; 12h; 16h post dose, on Day 2: 24h post dose, on Day 3: 1hr prior the second dose administration, on Days 4, 5, 6, 8, 10, 12, 13, 14: 1hr prior dosing, on Day 15 (last time the drug is administered): 1hr predose; 0,25h; 0,5h; 1h; 1,5h; 2h; 3h; 4h; 6h; 8h; 12h; 16h post dose, on Day 16: 24h post dose and Day 17: 48h post dose. This outcome measure shows the mean of all subject values resulting from each time point specified above.
PK of LML134: The average steady state serum concentration during multiple dosing (Cav,ss) in Part 2 | Starting 1hour prior the first dose administration (Day 1) until 48hour after the last dose administration (Day 17)
  Serum samples will be collected on Day 1: 1hr predose; 0,25h; 0,5h; 1h; 1,5h; 2h; 3h; 4h; 6h; 8h; 12h; 16h post dose, on Day 2: 24h post dose, on Day 3: 1hr prior the second dose administration, on Days 4, 5, 6, 8, 10, 12, 13, 14: 1hr prior dosing, on Day 15 (last time the drug is administered): 1hr predose; 0,25h; 0,5h; 1h; 1,5h; 2h; 3h; 4h; 6h; 8h; 12h; 16h post dose, on Day 16: 24h post dose and Day 17: 48h post dose. This outcome measure shows the mean of all subject values resulting from each time point specified above.
PK of LML134: The effective half-life based on drug accumulation at steady state (T1/2,acc) in Part 2 | Starting 1hour prior the first dose administration (Day 1) until 48hour after the last dose administration (Day 17)
  Serum samples will be collected on Day 1: 1hr predose; 0,25h; 0,5h; 1h; 1,5h; 2h; 3h; 4h; 6h; 8h; 12h; 16h post dose, on Day 2: 24h post dose, on Day 3: 1hr prior the second dose administration, on Days 4, 5, 6, 8, 10, 12, 13, 14: 1hr prior dosing, on Day 15 (last time the drug is administered): 1hr predose; 0,25h; 0,5h; 1h; 1,5h; 2h; 3h; 4h; 6h; 8h; 12h; 16h post dose, on Day 16: 24h post dose and Day 17: 48h post dose. This outcome measure shows the mean of all subject values resulting from each time point specified above.
PK of LML134: The accumulation ratio (Racc) in Part 2 | Starting 1hour prior the first dose administration (Day 1) until 48hour after the last dose administration (Day 17)
  Serum samples will be collected on Day 1: 1hr predose; 0,25h; 0,5h; 1h; 1,5h; 2h; 3h; 4h; 6h; 8h; 12h; 16h post dose, on Day 2: 24h post dose, on Day 3: 1hr prior the second dose administration, on Days 4, 5, 6, 8, 10, 12, 13, 14: 1hr prior dosing, on Day 15 (last time the drug is administered): 1hr predose; 0,25h; 0,5h; 1h; 1,5h; 2h; 3h; 4h; 6h; 8h; 12h; 16h post dose, on Day 16: 24h post dose and Day 17: 48h post dose. This outcome measure shows the mean of all subject values resulting from each time point specified above.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Novartis Pharmceuticals
Locations (1):
- Novartis Investigative Site, Berlin, Germany